CLINICAL TRIAL: NCT02317367
Title: Self-Affirmation: Construct Validity
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999915032; 15-C-N032
Record Dates: First submitted 2014-12-13; First posted 2014-12-16 (Estimated); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Risk Reduction Behavior
Keywords: Construct Validity; Self-Affirmation; Alcohol Consumption; Breast Cancer
MeSH Terms: conditions — Risk Reduction Behavior; Alcohol Drinking; Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- adult women: Women who drink seven or more drinks per week
- adults a: Individuals who eat fewer than five servings of fruits and vegetables per day, on average, based on an NCI screener for fruit and vegetable consumption.
- adults b: Individuals who exercise (moderate or vigorous intensity) less than 75 minutes per week.

SUMMARY:
Background:

- People respond differently when asked about their values. They also respond differently when they learn about how their actions affect their lives and health. Researchers want to learn more about these differences. This can help them improve public health messages.

Objective:

- To see how people respond differently to questions about their values and to information about alcohol and breast cancer.

Eligibility:

Study 1

- Women age 18 and older.

Study 2 & Study 3

-Women and men aged 18 and older to take part in these studies if they do not meet the US recommendations of eating 5 or more servings of fruits and vegetables per week.

Design:

* This study will take place online.
* Participants will be randomly assigned to a group that will complete a certain task.
* Researchers will ask participants to complete 2 small studies:
* Values Study. Some participants may write briefly about a value that is important to them or to someone they are close to. Some participants will complete a short questionnaire instead of the writing exercise.
* Study 1:

Alcohol and Breast Cancer Study. Participants will read a health message. This will be about the link between alcohol use and increased breast cancer risk. Participants will then answer questions about what they read and their beliefs about alcohol and breast cancer.

-Study 2:

Fruit and Vegetable Consumption and Health Study. Participants will read a health message about the fruit and vegetable consumption. Participants will then answer questions about what they read and their beliefs about fruit and vegetable consumption.

-Study 3:

Fruit and Vegetable Consumption and Health Study. Participants will read a health message about the fruit and vegetable consumption. Participants will then answer questions about what they read and their beliefs about fruit and vegetable consumption. Complete a follow-up survey that will be emailed to you through the mTurk system a week after you complete the main study.

* Both studies in either Study 1, Study 2 and Study 3 should take about 30 minutes.

DETAILED DESCRIPTION:
Self-affirmation, a process by which individuals reflect on cherished personal values is a potent means of augmenting the effectiveness of threatening health communications. Individuals tend to be defensive against information suggesting their behavior puts them at risk for disease or negative health. Previous evidence suggests that self-affirmation may reduce defensiveness to threatening health information, increasing openness to the message and resulting in increased disease risk perceptions, disease-related worry, intentions to engage in preventive behavior, and actual behavioral change. Understanding the mechanisms that explain these robust effects would yield evidence important for dissemination, including ways to refine self-affirmation interventions and make them more potent, which could change the ways that public health messages are constructed. Thus, we aim to elucidate potential mechanisms underlying the effectiveness of self-affirmation, including self-activation, general affirmation, and domain-specific affirmation. In study 1, female human subjects will be randomly assigned to one of eleven affirmation or self- activation conditions. Following the affirmation or activation task, subjects will read about the documented link between alcohol and breast cancer. Finally, they will be asked a series of questions about their intentions to reduce drinking, their perceived risk of breast cancer, and their worry about breast cancer. Study 2 will replicate study 1, but in a different behavioral domain (physical activity) and a different sample (both males and females who do not meet physical activity recommendations). Study 3 will extend Studies 1 and 2 by examining whether the most effective self-affirmations identified in these studies produce short-term increases in fruit and vegetable consumption. Drawing on previous research, we hypothesize these inductions will be effective to the degree that they involve a self-affirmation, but will not be effective if they involve only other-affirmation or self-activation.

ELIGIBILITY:
* INCLUSION CRITERIA:

Study 1:

Amazon mTurk workers will be invited to participate if they are women over the age of 18. They will also be screened to meet alcohol consumption inclusion criteria. Women will be eligible to complete the study if they drink seven or more drinks per week (consistent with the alcohol consumption level the health message links to increased breast cancer risk (which is based on evidence in the extant breast cancer risk literature). If women report drinking 7 or more drinks in a sitting, they will be eligible regardless of how many times they drank in the past year. If they report drinking less than 7 drinks in a sitting, an average will be calculated to determine whether they meet inclusion criteria. For example, women who report drinking twice per week on average, and who drink an average of 4 drinks in a sitting, would be eligible for the study.

Study 2:

Prolific participants will be invited to take part in the study if they are over the age of 18. They will also be screened to meet fruit and vegetable consumption inclusion criteria. Individuals will be eligible to complete the study if they eat fewer than 5 servings of fruits and vegetables per day, on average (consistent with the consumption level the health message, and consistent with US consumption recommendations).

Study 3:

Amazon mTurk workers will be invited to participate if they are over the age of 18. They will also be screened to meet fruit and vegetable consumption inclusion criteria. Individuals will be eligible to complete the study if they eat fewer than 5 servings of fruits and vegetables per day, on average (consistent with the consumption level the health message, and consistent with US consumption recommendations).

EXCLUSION CRITERIA:

Study1

All men, and women who report a lower threshold of alcohol consumption, will be excluded.

Study 2

All individuals who report a higher threshold of physical activity will be excluded

Study3

All individuals who report a higher threshold of fruit and vegetable. consumption, will be excluded. All individuals who participated in Studies 1 and 2 will be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Convenience sample of online panelists in Amazon's mTurk pool (female alcohol drinkers only for study 1; guidelines/fruit and vegetable consumption guidelines for study 3).Convenience sample of online panelists in Prolific's pool (males and females who do not meet physical activity for Study 2)
Sampling Method: Non-Probability Sample
Enrollment: 3112 (Actual)
Dates: Start 2016-07-31 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
Intentions to reduce alcohol consumption | Immediately post-intervention
  Intentions to reduce alcohol consumption
Intentions to increase physical activity | immediately post-intervention
  Intentions to increase physical activity

CONTACTS AND LOCATIONS:
Overall Officials: William M Klein, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Crocker J, Niiya Y, Mischkowski D. Why does writing about important values reduce defensiveness? Self-affirmation and the role of positive other-directed feelings. Psychol Sci. 2008 Jul;19(7):740-7. doi: 10.1111/j.1467-9280.2008.02150.x. PMID 18727791